CLINICAL TRIAL: NCT06931002
Title: Human Bronchiectasis Rhinovirus Challenge to Define Immunopathogenesis of Exacerbation
Brief Title: A Rhinovirus Challenge Study to Investigate Exacerbations and Immune Responses in Bronchiectasis
Acronym: BARRIER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23IC8574
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Bronchiectasis Adult; Bronchiectasis With Acute Exacerbation; Bronchiectasis With Chronic Infection With Pseudomonas Aeruginosa; Viral Infection; Rhinovirus Infection
Keywords: bronchiectasis; rhinovirus; case control study
MeSH Terms: conditions — Virus Diseases; Bronchiectasis

STUDY DESIGN:
Intervention Model Description: All participants in the study will be challenged with Rhinovirus A16.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rhinovirus Challenge (Other): All patients in the study will receive Rhinovirus A-16
  Interventions: Biological: Rhinovirus A-16 Infection

INTERVENTIONS:
Biological: Rhinovirus A-16 Infection — All participants will be deliberately infected with Rhinovirus A-16

SUMMARY:
The goal of this study is to determine if viral infection with the common cold leads to an exacerbation in participants with bronchiectasis. The investigators will compare the participants with bronchiectasis to a group of healthy participants. The main questions it aims to answer are:

* Does viral infection with the common cold lead to an exacerbation in bronchiectasis?
* Does the immune response differ to that of a healthy participant?

Participants will attend for a screening visit to see if they are eligible. All participants who are eligible and have consented to take part will have baseline investigations done including blood tests and a bronchoscopy. They will be given a spray of a virus that causes the common cold into their nose. They will then be followed up over the next 6 weeks with some of the following procedures at each study visit; spirometry, nasosorption, nasal lavage, nasal brushing, blood test, sputum collection and a bronchoscopy. Participants will be asked to keep a daily record of their symptoms throughout the study.

DETAILED DESCRIPTION:
Study Rationale:

Bronchiectasis is a chronic respiratory disease affective >200,000 individuals in the UK. The investigators are aiming to develop an experimental rhinovirus challenge model for bronchiectasis. This model could provide crucial insights into how viral infections trigger exacerbations (flare-ups) in bronchiectasis patients. Recent studies have found that viruses, especially rhinoviruses, are present in a significant number of bronchiectasis exacerbations. However, their exact role and the mechanisms behind increased viral susceptibility in these patients remain unclear. This model will allow us to study how factors like altered lung microbiota, might influence viral susceptibility. By enabling controlled sampling of both upper and lower airways at specific times during an infection, this study offers a opportunity to understand the complex immunological responses involved. Currently there is a poor understanding of exacerbation mechanisms in bronchiectasis and future development of treatment strategies require a suitable translational system for testing. This research could shed light on why bronchiectasis patients are more vulnerable to viral infections and potentially pave the way for new strategies to predict, prevent, or manage exacerbations.

End of Study:

• Follow-up period of 42 days.

Study Centres:

• There will be 1 study centre, ICRRU within Imperial College Healthcare NHS site at St Mary's Hospital London, United Kingdom.

Study Intervention:

• All participants will be inoculated intra-nasally with rhinovirus A-16.

Study Procedures:

* Screening period (lung function tests (FEV1, FVC and PEF), height and weight/BMI, Medical and surgical history, drug history, pregnancy test for females, Lung function tests (FEV1, FVC, PEF), blood sample, nasosorption and nasal brushing.
* Baseline visit to clinic (Blood tests including for haematology, biochemistry and coagulation), vital signs, physical examination, nasosorption, nasal brushings, spontaneous sputum collection, chest x-ray, lung function tests (FEV1, FVC, PEF and FeNO) and a stool sample.
* Baseline bronchoscopy: (Blood tests, nasosorption, nasal brushings and bronchoscopy including bronchoabsorption, bronchioalveolar lavage, bronchial brushings and bronchial biopsies)
* Viral inoculation: (Vital signs, physical examination, nasal lavage, spontaneous sputum collection and intranasal RV-A16 challenge)
* Visit Day 1: (Vital signs, physical examination, review of symptom scores, nasosorption, nasal lavage, nasal brushing, spontaneous sputum collection and lung function tests (FEV1, FVC and PEF))
* Visit Day 2: (Vital signs, physical examination, review of symptom scores, bloods, nasal lavage, spontaneous sputum collection and lung function tests (FEV1, FVC and PEF))
* Visit Day 4: (Vital signs, physical examination, review of symptom scores, nasal lavage, spontaneous sputum collection and lung function tests (FEV1, FVC and PEF))
* Visit Day 7 and Bronchoscopy: (Vital signs, physical examination, review of symptom scores, blood tests, nasosorption, nasal lavage, nasal brushings, lung function tests (FEV1, FVC, PEF and FeNO), stool sample and bronchoscopy including bronchoabsorption, bronchioalveolar lavage, bronchial brushings and bronchial biopsies)
* Visit Day 10: (Vital signs, physical examination, review of symptom scores, nasal lavage, spontaneous sputum collection and lung function tests (FEV1, FVC and PEF))
* Visit Day 14: (Vital signs, physical examination, review of symptom scores, bloods, nasosorption, nasal lavage, spontaneous sputum collection and lung function tests (FEV1, FVC and PEF))
* Visit Day 21: (Vital signs, physical examination, review of symptom scores, nasal lavage, spontaneous sputum collection and lung function tests (FEV1, FVC and PEF))
* Visit Day 28: (Vital signs, physical examination, review of symptom scores, nasal lavage, spontaneous sputum collection and lung function tests (FEV1, FVC and PEF))
* Visit Day 42: (Vital signs, physical examination, review of symptom scores, bloods, nasosorption, nasal lavage, nasal brush, spontaneous sputum collection and lung function tests (FEV1, FVC and PEF) and stool sample)

Study Sample Size:

• 18 participants will be recruited with bronchiectasis, 18 patients with bronchiectasis and chronic pseudomonas colonisation and 18 healthy participants will be recruited.

Statistical Methods:

• Using an independent two-sided t-test a sample size of 15 participants per group will allow the detection of a significant difference in lower respiratory tract symptom scores and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* For healthy volunteers:

  1) Age 18 to 65 years.
* For bronchiectasis study subjects:

  1. Confirmed diagnosis of bronchiectasis aged 18-65 years with bronchiectasis severity index score of 0-8 .
  2. For Pseudomonas colonised individuals, isolation of Pseudomonas aeruginosa in two or more cultures, at least 3 months apart in a 2-year period.

Exclusion Criteria:

* For healthy volunteers and bronchiectasis study subjects:

  1. Any medical co-morbidity impacting the study in the opinion of the medical team
  2. Current smoking history within last 12 months or ex smoking history >5 pack years
  3. Pre-existing serum neutralising antibodies to RV-A16 (strain to be used for challenge)
  4. Close contact with infants or elderly individuals either at home or workplace
  5. Pregnancy or breastfeeding
* For bronchiectasis study subjects:

  1) Individuals with bronchiectasis secondary to cystic fibrosis, primary immunodeficiency, primary ciliary dyskinesia and allergic bronchopulmonary aspergillosis 2) Individuals with other significant chronic lung disease diagnoses (eg. interstitial lung disease) which would impact the study in the opinion of the medical team 4) FEV1 < 50% predicted 8) Recent antibiotics for exacerbations within the preceding 6 weeks and prophylactic antibiotics (azithromycin or nebulised antibiotics) within preceding 4 weeks 9) Corticosteroid use (inhaled, nasal or systemic) within preceding 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Lower respiratory tract symptom scores | From enrolment to the end of the study at 42 days post viral innoculation
  Participants will be asked to record their lower respiratory tract symptom scores daily at prior to and in the 42 days following viral infection with rhinovirus A-16. Participants will rate their shortness of breath, and wheeze on a scale of 0 to 4, with 0 being no symptoms at all and 4 being symptoms at rest. They will rate their cough on a scale of 0 to 3, 0 being no cough and 3 being a severe cough. They will rate their sputum quantity on a scale from 0 to 3, with 0 being no sputum and 3 being large volumes of sputum (>100ml). They will also rate their sputum quality on a score from 0 to 3, with 0 being no sputum and 3 being purulent (green) sputum.

SECONDARY OUTCOMES:
Sputum Viral Load | From day 1 post viral innoculation to day 42.
  The investigators will use qPCR to measure viral load in spontaneously expectorated sputum produced by patients at study visits.
Sputum Neutrophils | From day 1 post viral inoculation to day 42.
  The investigators will use flow cytometry to measure sputum neutrophils on spontaneously expectorated sputum from day 1 to day 42.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Shah, PhD, Principal Investigator — Imperial College London; Aran Singanayagam, PhD, Principal Investigator — Imperial College London; Sebastian Johnston, PhD, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital - Imperial Clinical Respiratory Research Unit (ICRRU), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The investigators will not be sharing individual participant data to protect patient confidentiality and privacy.

REFERENCES:
- See also: Website providing information about the study — https://www.imperial.ac.uk/infectious-disease/research/human-challenge/barrier-study/